CLINICAL TRIAL: NCT01266720
Title: Phase 1 Study of HLA-A*0201 Restricted Antiangiogenic Peptide Vaccine Therapy Using Epitope Peptide Derived From VEGFR1 and VEGFR2 With Gemcitabine in Treating Patients With Unresectable, Recurrent, or Metastatic Pancreatic Cancer
Brief Title: HLA-A*0201 Restricted Peptide Vaccine Therapy With Gemcitabine With Gemcitabine in Patient Pancreatic Cancer (Phase1)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fukushima Medical University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Fukushima Medical University (Department of Regeneration Surgery), Fukushima Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 689
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-12

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; peptide vaccine; VEGFR; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Receptor Protein-Tyrosine Kinases; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase 1 study (Experimental): Interventions:
  Biological: VEGFR1, VEGFR2 Drug: Gemcitabine
  Interventions: Biological: VEGFR1, VEGFR2; Drug: Gemcitabine

INTERVENTIONS:
Biological: VEGFR1, VEGFR2 — One mg of each peptide will be administered subctaneously on days 1, 8, 15 and 22
  Other Names: VEGFR1 and VEGFR2 specific epitope vaccine
Drug: Gemcitabine — Gemcitabine will be administered intravenously at a fixed dose of 1000mg/m2 on day 1, 8, 15.
  Other Names: Gemzar

SUMMARY:
The purpuse of this study is to assess toxicities of angiogenic peptide vaccine therapy with gemcitabine in treating HLA-A*0201 restricted patient with non-resectable pancreatic cancer.

DETAILED DESCRIPTION:
The prognosis of pancreatic cancer is extremely poor even with extensive surgery, chemotherapy or radiation. It has been required development of new treatment modalities. Immunotherapy is one of the encouraging modalities for cancer patients. The investigators have to assess its toxicities and immune responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic pancreatic cancer precluding curative surgical resection and recurrent pancreatic cancer
* Measurable disease by CT scan
* ECOG performance status 0-2
* Life expectancy > 3 months
* laboratory values as follows: 2,000/mm3 < WBC < 15,000/mm3, Platelet count >75,000/mm3, Total Bilirubin <1.5 mg/dl, Asparate transaminase <150IU/L, Alanine transaminase < 150 IU/L, Creatinine < 3.0mg/dl
* HLA-A*0201
* Able and willing to give valid written infromed consent

Exclusion Criteria:

* Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
* Breast-feeder
* Active or uncontrolled infection
* Prior chemotherapy, radiation therapy, or immunotherapy within 4 weeks
* Serious or uncured wound
* Active or uncontrolled other malignancy
* Steroids or immunosuppressing agent dependent status
* Interstitial pneumonia
* Ileus
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Toxicities as assessed by NCI-CACAE ver3 | 3 months

SECONDARY OUTCOMES:
Differences of peptide specific CTL response in vitro among sequence of gemcitabine and peptide vaccine administration | 3 months
CD8 population | 3 months
Change in level of regulatory T cells | 3 months
Objective response rate | 1 year
Feasibility | 1 year
Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mitsukazu Gotoh, MD & PhD, Study Chair — Fukushima Medical University, Department of Regeneration Surgery
Locations (1):
- Fukushima Medical University Hospital, Fukushima, Fukushima, Japan

REFERENCES:
- [Background] Niethammer AG, Xiang R, Becker JC, Wodrich H, Pertl U, Karsten G, Eliceiri BP, Reisfeld RA. A DNA vaccine against VEGF receptor 2 prevents effective angiogenesis and inhibits tumor growth. Nat Med. 2002 Dec;8(12):1369-75. doi: 10.1038/nm1202-794. Epub 2002 Nov 4. PMID 12415261
- [Background] Ishizaki H, Tsunoda T, Wada S, Yamauchi M, Shibuya M, Tahara H. Inhibition of tumor growth with antiangiogenic cancer vaccine using epitope peptides derived from human vascular endothelial growth factor receptor 1. Clin Cancer Res. 2006 Oct 1;12(19):5841-9. doi: 10.1158/1078-0432.CCR-06-0750. PMID 17020992
- [Background] Wada S, Tsunoda T, Baba T, Primus FJ, Kuwano H, Shibuya M, Tahara H. Rationale for antiangiogenic cancer therapy with vaccination using epitope peptides derived from human vascular endothelial growth factor receptor 2. Cancer Res. 2005 Jun 1;65(11):4939-46. doi: 10.1158/0008-5472.CAN-04-3759. PMID 15930316